CLINICAL TRIAL: NCT04550234
Title: A Randomised, Single Dose, 5-period, 5-treatment, Crossover Study to Assess the Relative Bioavailability of 4 Different Formulations of Verinurad and Allopurinol in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Assess Drug Availability of 4 Different Formulations of Verinurad and Allopurinol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5495C00014
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease
Keywords: 3-period; Crossover; URAT1 inhibitor; Xanthine oxidase inhibitor
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Allopurinol; verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment 1 (Experimental): Subjects will receive verinurad prolonged release HPMC capsule and allopurinol tablet in fasted state on Day 1.
  Interventions: Drug: Verinurad prolonged release HPMC capsule; Drug: Allopurinol Tablet
- Treatment 2 (Experimental): Subjects will receive verinurad/allopurinol FDC capsule in fasted state on Day 1.
  Interventions: Drug: Verinurad/Allopurinol FDC Capsule
- Treatment 3 (Experimental): Subjects will receive verinurad/allopurinol FDC capsule in fed state on Day 1.
  Interventions: Drug: Verinurad/Allopurinol FDC Capsule
- Treatment 4 (Experimental): Subjects will receive verinurad prolonged release HPMC capsule and allopurinol tablet in fed state on Day 1.
  Interventions: Drug: Verinurad prolonged release HPMC capsule; Drug: Allopurinol Tablet
- Treatment 5 (Experimental): Subjects will receive verinurad prolonged release gelatin capsule in fasted state on Day 1.
  Interventions: Drug: Verinurad prolonged release gelatin Capsule

INTERVENTIONS:
Drug: Verinurad prolonged release HPMC capsule — Randomized subjects will receive oral dose of verinurad HPMC capsule.
  Arms: Treatment 1; Treatment 4
Drug: Allopurinol Tablet — Randomized subjects will receive oral dose of allopurinol tablet.
  Arms: Treatment 1; Treatment 4
Drug: Verinurad/Allopurinol FDC Capsule — Randomized subjects will receive oral dose of Verinurad/Allopurinol FDC capsule.
  Arms: Treatment 2; Treatment 3
Drug: Verinurad prolonged release gelatin Capsule — Randomized subjects will receive oral dose of Verinurad gelatin capsule.
  Arms: Treatment 5

SUMMARY:
This study is a single centre, randomised, open-label, single-dose, 5-period, 5-treatment, crossover study in healthy male and female subjects. This study is intended to assess the relative bioavailability between the fixed dose combination (FDC, i.e. verinurad/allopurinol FDC capsule 12/300 mg) and free combination formulations of verinurad (i.e. verinurad prolonged release Hydroxypropyl methylcellulose [HPMC] capsule 12 mg) and allopurinol (i.e. allopurinol table 300 mg) in fasted and fed conditions. The study will also assess the relative bioavailability between a formulation only containing verinurad (i.e. verinurad prolonged release gelatin capsule 12 mg) and the FDC capsule.

DETAILED DESCRIPTION:
The study comprises of:

* A Screening Period of maximum 28 days;
* Five treatment periods during which subjects will be resident from the morning of Day -2 until at least 72 hours after dosing in Treatment Period 5; discharged on the morning of Day 4 of Treatment Period 5; and
* A Follow-up Visit 7 to 14 days after the last dosing.

Each subject will receive 5 single dose treatments of verinurad and allopurinol or verinurad alone and subject will be involved in the study for 52 to 59 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venepuncture.
* Have a body mass index between 18 and 30 kg/m^2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).
* Females must have a negative pregnancy test at screening and on admission to the unit and must be:

  1. not pregnant or currently lactating or breastfeeding.
  2. of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria: (i) postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the postmenopausal range (FSH levels > 40 IU/mL).

     (ii) documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
  3. OR if of childbearing potential must be willing to use an acceptable method of contraception to avoid pregnancy for the entire study period.
* Must be able to swallow multiple capsules and tablets.

Exclusion Criteria:

* History of gout or any clinically significant disease which, in the opinion of the principal investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of verinurad.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results as judged by the Investigator at screening and first admission, including:

  1. Alanine aminotransferase > 1.5 x upper limit of normal (ULN),
  2. Aspartate aminotransferase > 1.5 x ULN,
  3. Bilirubin (total) > 1.5 x ULN,
  4. Gamma glutamyl transpeptidase > 1.5 x ULN.
* Any clinically significant abnormal findings in vital signs at the Screening Visit and/or admission to the Clinical Unit, including, but not limited to, any of the following:

  1. Pulse (resting, supine) < 50 beats per minute (bpm) or > 90 bpm,
  2. Systolic blood pressure (BP) < 90 mmHg or > 140 mmHg and/or diastolic BP < 50 mmHg or > 90 mmHg sustained for > 10 minutes while resting in a supine position.
* Any clinically significant abnormalities on 12 lead electrocardiogram (ECG) at the Screening Visit, including, but not limited to any of the following:

  1. QTcF > 450 ms or < 340 ms or family history of long QT syndrome,
  2. Any significant arrhythmia
  3. Conduction abnormalities
  4. Clinically significant PR (PQ) interval prolongation (> 240 ms); intermittent second or third degree AV block, or AV dissociation
  5. Complete bundle branch block and/or QRS duration > 120 ms.
* Any positive result at the Screening Visit for serum Hepatitis B surface antigen or Anti Hepatitis B core antibody, hepatitis virus C antibody, and human immunodeficiency virus antibody.
* Suspicion or known Gilbert's and/or Lesch Nyhan syndrome.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
* Has received another new chemical or biological entity within 30 days or at least 5 half lives of the first administration of verinurad in this study.
* Subjects who have previously received verinurad.
* Plasma donation within 1 month of screening or any blood donation/loss of more than 500 mL during the 3 months prior to the Screening Visit.
* Subjects who are pregnant, lactating or planning to become pregnant.
* Hypersensitivity to verinurad, allopurinol or any drug with a similar chemical structure/class to verinurad and/or allopurinol.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.
* Excessive intake of caffeine containing drinks or food as judged by the PI.
* Positive screen for drugs of abuse or cotinine (nicotine) at the Screening Visit or positive screen for alcohol, drugs of abuse and cotinine on each admission to the study centre.
* Use of drugs with enzyme inducing properties within 3 weeks prior to the first administration of verinurad.
* Use of any prescribed or non prescribed medication including antacids, analgesics, herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of verinurad or longer if the medication has a long half life.
* Any AstraZeneca, Parexel or study site employee or their close relatives.
* Subjects who cannot communicate reliably with the PI and/or is not able to read, speak and understand the German language.
* Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Subjects with any special dietary restrictions such as subjects that are lactose intolerant or are vegetarians/vegans.
* Subject is a carrier of the HLA B*58:01 allele.
* Subject has a positive test result for severe acute respiratory syndrome corona virus (SARS-CoV-2) RT-PCR before randomisation.
* Subject has clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19), eg, fever, dry cough, dyspnoea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* History of severe COVID-19 (hospitalisation, extracorporeal membrane oxygenation, mechanically ventilated).
* Subjects who are regularly exposed to COVID-19 as part of their daily life.
* Subjects who have had or are planning to have the COVID-19 vaccination within 4 weeks prior to screening or at any time during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the requests portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D5495C00014 CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00014&attachmentIdentifier=5bd8c3ee-4ea2-4d8c-833e-9e108efe7d44&fileName=D5495C00014_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D5495C00014 Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00014&attachmentIdentifier=505ef90d-887e-4b32-8472-68345ad56b7a&fileName=D5495C00014_Final_Protocol_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 13 April 2021 to 15 July 2021.
Pre-assignment Details: Subjects who met all the inclusion and none of the exclusion criteria were randomized at single center. The screening period was from Day -28 to Day -3. Informed consent form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment.
Groups:
- Treatment Sequence 12345: Subjects received single-dose treatments of verinurad and allopurinol or verinurad alone on 5 occasions [Treatment 1: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fasted state; Treatment 2: verinurad/allopurinol FDC capsule, fasted state; Treatment 3: verinurad/allopurinol FDC capsule, fed state; Treatment 4: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fed state; Treatment 5: verinurad prolonged release gelatin capsule, fasted state] on Day 1 separated by at least 5 days washout between IMP administration.
- Treatment Sequence 23451: Subjects received single-dose treatments of verinurad and allopurinol or verinurad alone on 5 occasions [Treatment 2: verinurad/allopurinol FDC capsule, fasted state; Treatment 3: verinurad/allopurinol FDC capsule, fed state; Treatment 4: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fed state; Treatment 5: verinurad prolonged release gelatin capsule, fasted state; Treatment 1: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fasted state] on Day 1 separated by at least 5 days washout between IMP administration.
- Treatment Sequence 34512; Treatment Sequence 45123: Subjects received single-dose treatments of verinurad and allopurinol or verinurad alone on 5 occasions [Treatment 3: verinurad/allopurinol FDC capsule, fed state; Treatment 4: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fed state; Treatment 5: verinurad prolonged release gelatin capsule, fasted state; Treatment 1: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fasted state; Treatment 2: verinurad/allopurinol FDC capsule, fasted state] on Day 1 separated by at least 5 days washout between IMP administration.
- Treatment Sequence 51234: Subjects received single-dose treatments of verinurad and allopurinol or verinurad alone on 5 occasions [Treatment 5: verinurad prolonged release gelatin capsule, fasted state; Treatment 1: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fasted state; Treatment 2: verinurad/allopurinol FDC capsule, fasted state; Treatment 3: verinurad/allopurinol FDC capsule, fed state; Treatment 4: verinurad prolonged release HPMC capsule and allopurinol tablet, as a free combination, fed state] on Day 1 separated by at least 5 days washout between IMP administration.
Period: Overall Study
Arm/Group | Treatment Sequence 12345 | Treatment Sequence 23451 | Treatment Sequence 34512 | Treatment Sequence 45123 | Treatment Sequence 51234
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set consisted of all subjects randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 12345 | Treatment Sequence 23451 | Treatment Sequence 34512 | Treatment Sequence 45123 | Treatment Sequence 51234 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (7.4) | 34.2 (8.0) | 26.0 (5.0) | 33.0 (4.7) | 38.4 (10.6) | 32.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 5 | 2 | 13
  Male | 2 | 4 | 3 | 0 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 4 | 4 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 5 | 5 | 5 | 22
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Cmax: Maximum Observed Plasma Drug Concentration
Description: The Cmax of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: The PK analysis set included all subjects in the safety analysis set who received a verinurad + allopurinol (or verinurad alone for Treatment 5) dose and who had at least one quantifiable post-dose plasma concentration.
  Here, number analysed in each row signifies the subjects with available data that were analysed for each drug for that outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre
Groups:
- Treatment 1: Subjects received verinurad prolonged release HPMC capsule and allopurinol tablet as a free combination in fasted state on Day 1
- Treatment 2: Subjects received verinurad/allopurinol FDC capsule in fasted state on Day 1
- Treatment 3: Subjects received verinurad/allopurinol FDC capsule in fed state on Day 1
- Treatment 4: Subjects received verinurad prolonged release HPMC capsule and allopurinol tablet in fed state on Day 1
- Treatment 5: Subjects received verinurad prolonged release gelatin capsule in fasted state on Day 1
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
nanogram/millilitre
  Verinurad | 26.62 (50.71) | 34.95 (61.87) | 20.18 (70.96) | 13.86 (68.98) | 35.35 (44.84)
  Allopurinol | 1526 (37.98) | 1471 (42.92) | 1079 (68.87) | 1627 (43.71) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 6376 (16.67) | 6066 (21.61) | 5269 (19.91) | 5709 (21.21) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
Statistical Analysis 1: Comparison: Treatment 2 vs Treatment 3; Statistical Comparison of Verinurad Analysis of variance (ANOVA) of log transformed PK parameter with treatment, sequence, period as fixed effects and subject nested within sequence as random effect; Test type: Other; Geometric mean ratio = 57.73, 90% CI 2-sided [47.07 to 70.81]
Statistical Analysis 2: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 145.55, 90% CI 2-sided [118.66 to 178.52]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 52.07, 90% CI 2-sided [42.46 to 63.87]
Statistical Analysis 4: Comparison: Treatment 2 vs Treatment 5; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 101.16, 90% CI 2-sided [82.48 to 124.08]
Statistical Analysis 5: Comparison: Treatment 2 vs Treatment 3; Statistical Comparison of Allopurinol Analysis of variance (ANOVA) of log transformed PK parameter with treatment, sequence, period as fixed effects and subject nested within sequence as random effect; Test type: Other; Geometric mean ratio = 73.34, 90% CI 2-sided [61.81 to 87.03]
Statistical Analysis 6: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 66.33, 90% CI 2-sided [55.90 to 78.72]
Statistical Analysis 7: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 106.58, 90% CI 2-sided [89.81 to 126.47]
Statistical Analysis 8: Comparison: Treatment 2 vs Treatment 3; Statistical Comparison of Oxypurinol Analysis of variance (ANOVA) of log transformed PK parameter with treatment, sequence, period as fixed effects and subject nested within sequence as random effect; Test type: Other; Geometric mean ratio = 86.86, 90% CI 2-sided [83.15 to 90.74]
Statistical Analysis 9: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 92.30, 90% CI 2-sided [88.35 to 96.42]
Statistical Analysis 10: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 89.54, 90% CI 2-sided [85.71 to 93.54]

2. Secondary Outcome: AUCinf: Area Under Plasma Concentration-time Curve From 0 to Infinity
Description: The AUCinf of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/millilitre
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour*nanogram/millilitre
  Verinurad | 180.4 (48.87) | 195.2 (48.63) | 200.1 (54.89) | 138.4 (64.06) | 187.8 (40.22)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 4486 (37.86) | 4332 (46.40) | 3551 (37.17) | 4114 (35.79) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 170100 (19.07) | 167900 (24.10) | 153200 (24.22) | 153300 (22.74) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
Statistical Analysis 1: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 102.49, 90% CI 2-sided [89.12 to 117.86]
Statistical Analysis 2: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 144.61, 90% CI 2-sided [125.75 to 166.31]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 76.72, 90% CI 2-sided [66.71 to 88.23]
Statistical Analysis 4: Comparison: Treatment 2 vs Treatment 5; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 96.19, 90% CI 2-sided [83.64 to 110.62]
Statistical Analysis 5: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 89.41, 90% CI 2-sided [83.86 to 95.34]
Statistical Analysis 6: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 94.16, 90% CI 2-sided [88.31 to 100.40]
Statistical Analysis 7: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 91.70, 90% CI 2-sided [86.37 to 97.36]
Statistical Analysis 8: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 91.23, 90% CI 2-sided [88.01 to 94.56]
Statistical Analysis 9: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 99.95, 90% CI 2-sided [96.43 to 103.61]
Statistical Analysis 10: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 90.13, 90% CI 2-sided [86.95 to 93.42]

3. Secondary Outcome: AUClast: Area Under Plasma Concentration-time Curve From Zero to the Last Quantifiable Concentration
Description: The AUClast of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour*nanogram/milliliter
  Verinurad | 169.3 (47.82) | 185.0 (49.64) | 190.3 (55.76) | 129.9 (65.65) | 176.4 (39.80)
  Allopurinol | 4407 (37.98) | 4251 (46.91) | 3512 (45.13) | 4030 (35.80) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 157100 (16.84) | 153100 (21.35) | 139200 (21.05) | 140100 (19.57) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
Statistical Analysis 1: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 102.91, 90% CI 2-sided [89.04 to 118.93]
Statistical Analysis 2: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 146.57, 90% CI 2-sided [126.82 to 169.40]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 76.72, 90% CI 2-sided [66.38 to 88.67]
Statistical Analysis 4: Comparison: Treatment 2 vs Treatment 5; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 95.37, 90% CI 2-sided [82.52 to 110.23]
Statistical Analysis 5: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 82.60, 90% CI 2-sided [77.38 to 88.17]
Statistical Analysis 6: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 87.14, 90% CI 2-sided [81.63 to 93.01]
Statistical Analysis 7: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 91.45, 90% CI 2-sided [85.67 to 97.61]
Statistical Analysis 8: Comparison: Treatment 2 vs Treatment 3; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 90.91, 90% CI 2-sided [87.98 to 93.94]
Statistical Analysis 9: Comparison: Treatment 3 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 99.37, 90% CI 2-sided [96.17 to 102.68]
Statistical Analysis 10: Comparison: Treatment 1 vs Treatment 4; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 89.18, 90% CI 2-sided [86.30 to 92.15]

4. Secondary Outcome: Tmax: Time to Reach Maximum Observed Plasma Concentration Following Drug Administration
Description: The tmax of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour
  Verinurad | 5.00 [3.00 to 6.02] | 4.00 [2.00 to 5.08] | 9.98 [3.00 to 12.03] | 5.03 [4.00 to 10.02] | 4.00 [2.00 to 6.00]
  Allopurinol | 1.50 [0.50 to 3.02] | 1.50 [0.50 to 4.02] | 3.00 [0.50 to 10.00] | 1.50 [0.50 to 5.00] | NA [NA to NA] — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 4.00 [1.00 to 6.00] | 4.00 [2.12 to 8.02] | 6.02 [1.00 to 12.03] | 4.00 [0.52 to 10.02] | NA [NA to NA] — As, subjects received only verinurad, hence this is not applicable

5. Secondary Outcome: Tlag: Time Delay Between Drug Administration and First Observed Concentration in Plasma
Description: The tlag of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour
  Verinurad | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 1.00] | 1.00 [0.00 to 2.02] | 1.02 [0.00 to 2.00] | 0.00 [0.00 to 0.50]
  Allopurinol | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 1.00] | 1.02 [0.00 to 4.00] | 0.00 [0.00 to 1.02] | NA [NA to NA] — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00] | NA [NA to NA] — As, subjects received only verinurad, hence this is not applicable

6. Secondary Outcome: t½λz: Half-life Associated With Terminal Slope (λz) of Semi-logarithmic Concentration-time Curve
Description: The t½λz of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour
  Verinurad | 15.57 (53.19) | 14.17 (58.62) | 13.69 (57.74) | 13.77 (61.38) | 14.71 (61.15)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 1.164 (21.78) | 1.142 (19.13) | 1.696 (56.37) | 1.085 (24.91) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 19.06 (19.81) | 20.45 (22.87) | 20.14 (23.18) | 20.21 (23.00) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

7. Secondary Outcome: λz: Terminal Elimination Rate Constant
Description: The λz of verinurad, allopurinol and oxypurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
per hour
  Verinurad | 0.04437 (55.10) | 0.04876 (65.26) | 0.04957 (61.83) | 0.05063 (57.34) | 0.04651 (60.92)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 0.5951 (21.96) | 0.6065 (18.98) | 0.4075 (57.03) | 0.6384 (25.11) | NA (NA) — As, subjects received only verinurad, hence this is not applicable
  Oxypurinol | 0.03653 (19.58) | 0.03309 (24.22) | 0.03512 (23.12) | 0.03425 (24.67) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

8. Secondary Outcome: CL/F: Apparent Total Body Clearance of Drug Clearance of Drug From Plasma After Extravascular Administration
Description: The CL/F of verinurad and allopurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Liter/hour
  Verinurad | 66.54 (48.87) | 61.46 (48.63) | 59.97 (54.90) | 86.73 (64.06) | 63.90 (40.22)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 66.88 (37.85) | 69.25 (46.40) | 84.47 (37.17) | 72.93 (35.78) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

9. Secondary Outcome: MRTinf: Mean Residence Time of the Unchanged Drug in the Systemic Circulation From Zero to Infinity
Description: The MRTinf of verinurad and allopurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour
  Verinurad | 18.99 (41.94) | 15.28 (43.14) | 18.91 (40.50) | 18.19 (38.37) | 15.94 (52.27)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 2.629 (18.88) | 2.950 (23.30) | 4.626 (43.33) | 2.827 (37.87) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

10. Secondary Outcome: Vz/F: Apparent Volume of Distribution During Terminal Phase After Extravascular Administration
Description: The Vz/F of verinurad and allopurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Liter
  Verinurad | 1495 (62.63) | 1256 (69.76) | 1184 (74.23) | 1723 (89.59) | 1356 (55.95)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 112.4 (31.38) | 114.2 (42.56) | 206.7 (80.39) | 114.1 (31.60) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

11. Secondary Outcome: Vss/F: Apparent Volume of Distribution at Steady State Following Extravascular Administration
Description: The Vss/F of verinurad and allopurinol were assessed as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Liter
  Verinurad | 1264 (55.42) | 939.3 (62.63) | 1134 (65.96) | 1578 (76.33) | 1018 (50.97)
  Allopurinol: number analyzed (Participants) | 25 | 25 | 21 | 25 | 25
  Allopurinol | 175.8 (37.01) | 204.3 (38.33) | 390.7 (65.33) | 206.1 (45.73) | NA (NA) — As, subjects received only verinurad, hence this is not applicable

12. Secondary Outcome: Emax, CB: Maximum Percentage Change From Baseline (CB)
Description: The Emax, CB in serum uric acid (sUA) concentration (time-matched, Day -1) was assessed as PD parameter.
Time Frame: Day -1, Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: The PD analysis set consisted of all subjects in the safety analysis set who received at least one of the verinurad and allopurinol (or verinurad alone for Treatment 5) doses and who had at least one quantifiable time-matched sUA concentration.
  Here, number analysed in each row signifies the subjects with available data that were analysed for each drug for that outcome measure.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
percentage (%) | -50.44 (8.304) | -53.84 (9.947) | -56.63 (9.618) | -54.43 (8.895) | -38.15 (9.724)

13. Secondary Outcome: tEmax, CB: Time of Maximum Percentage CB Change From Baseline (CB)
Description: The tEmax, CB in serum uric acid (sUA) concentration (time-matched, Day -1) was assessed as PD parameter.
Time Frame: Day -1, Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 12
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hour | 8.00 [6.00 to 48.00] | 6.00 [6.00 to 48.00] | 12.00 [6.00 to 48.00] | 12.00 [8.00 to 12.00] | 12.00 [4.00 to 48.00]

14. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events
Description: The safety of single doses of verinurad and allopurinol were assessed
Time Frame: From screening (Day -28 to -3) until follow-up visit (7 to 14 days post final dose) (approximately 52 to 59 days)
Population: The safety analysis set included all subjects who received at least one dose of IMP and for whom any safety post-dose data were available.
  Here, number analysed in each row signifies the subjects with available data that were analysed for each drug for that outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Participants
  Any AE | 8 | 2 | 2 | 6 | 2
  Any SAE | 0 | 0 | 0 | 0 | 0
  Any SAE with outcome of death | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 0 | 0 | 0 | 0
  Any possibly related AE | 3 | 1 | 1 | 3 | 1
  Any possibly related SAE | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: AUCinf: Area Under Plasma Concentration-time Curve From 0 to Infinity in Fasted Condition
Description: The AUCinf of verinurad, allopurinol and oxypurinol were assessed in fasted state as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/millilitre
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 25 | 25
hour*nanogram/millilitre
  Verinurad | 180.4 (48.87) | 195.2 (48.63)
  Allopurinol | 4486 (37.86) | 4332 (46.40)
  Oxypurinol | 170100 (19.07) | 167900 (24.10)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 108.25, 90% CI 2-sided [94.13 to 124.49]
Statistical Analysis 2: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 96.57, 90% CI 2-sided [90.96 to 102.53]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 98.75, 90% CI 2-sided [95.27 to 102.36]

16. Primary Outcome: AUClast: Area Under Plasma Concentration-time Curve From Zero to the Last Quantifiable Concentration in Fasted Condition
Description: The AUClast of verinurad, allopurinol and oxypurinol were assessed in fasted condition as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 25 | 25
hour*nanogram/milliliter
  Verinurad | 169.3 (47.82) | 185.0 (49.64)
  Allopurinol | 4407 (37.98) | 4251 (46.91)
  Oxypurinol | 157100 (16.84) | 153100 (21.35)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 109.27, 90% CI 2-sided [94.55 to 126.29]
Statistical Analysis 2: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 96.47, 90% CI 2-sided [90.38 to 102.97]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 97.48, 90% CI 2-sided [94.34 to 100.73]

17. Primary Outcome: Cmax: Maximum Observed Plasma Drug Concentration in Fasted State
Description: The Cmax of verinurad, allopurinol and oxypurinol were assessed in fasted state as PK parameters
Time Frame: Day 1, Day 2, Day 3 and Day 4 of each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 25 | 25
nanogram/millilitre
  Verinurad | 26.62 (50.71) | 34.95 (61.87)
  Allopurinol | 1526 (37.98) | 1471 (42.92)
  Oxypurinol | 6376 (16.67) | 6066 (21.61)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean ratio = 131.28, 90% CI 2-sided [107.03 to 161.02]
Statistical Analysis 2: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 5]; Test type: Other; Geometric mean ratio = 96.39, 90% CI 2-sided [81.23 to 114.39]
Statistical Analysis 3: Comparison: Treatment 1 vs Treatment 2; [analysis description as in outcome 1, analysis 8]; Test type: Other; Geometric mean ratio = 95.15, 90% CI 2-sided [91.08 to 99.40]

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to -3) until follow-up visit (7 to 14 days post final dose) (approximately 52 to 59 days)
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 8/25 | 2/25 | 2/25 | 6/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (N=25) | Treatment 2 (N=25) | Treatment 3 (N=25) | Treatment 4 (N=25) | Treatment 5 (N=25)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04550234/Prot_SAP_000.pdf